CLINICAL TRIAL: NCT02808793
Title: A Phase 1, Single Ascending Dose and Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AK002 in Patients With Indolent Systemic Mastocytosis
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AK002
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allakos Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK002-001
Record Dates: First submitted 2016-06-16; First posted 2016-06-22 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Indolent Systemic Mastocytosis
Keywords: ISM; Mastocytosis; Indolent Mastocytosis
MeSH Terms: conditions — Mastocytosis, Systemic; Mastocytosis | interventions — AK002

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AK002 (Experimental): IV dose of AK002
  Interventions: Drug: AK002

INTERVENTIONS:
Drug: AK002

SUMMARY:
This is a Phase 1 study to investigate the safety and tolerability of AK002 in patients with indolent systemic mastocytosis (ISM).

ELIGIBILITY:
Inclusion Criteria:

1. Provided written informed consent
2. Male or female aged ≥18 and ≤65 years at the time of signing the informed consent form
3. Confirmed diagnosis of ISM based on World Health Organization (WHO) criteria (Appendix 1)
4. Presence of at least 1 of the following SM related symptoms:

   1. Flushing (at least 1 episode per week)
   2. Pruritus (minimum MAS2 score of 4) (Appendix 2)
   3. Diarrhea (minimum MAS2 score of 4) (Appendix 2)
   4. Anaphylaxis (at least 1 episode [grade 2 or higher] within the last 12 months)
5. Serum total tryptase exceeded 15 ng/mL* at 2 or more measurements obtained 1 or more months apart within the last 2 years (*Note: this varies from the minor criterion of "persistently exceeds 20 ng/mL" in the WHO criteria for diagnosis of ISM)
6. Willing and able to comply with the study procedures and visit schedule, including follow-up visits
7. Able to communicate effectively with the study site personnel
8. Negative Screening urine drug tests (alcohol, amphetamines/methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, cotinine, methadone, methaqualone, opiates, phencyclidine)
9. Negative Screening ova and parasite test
10. Determined by the Investigator to be in good health as documented by the medical history, physical examination (PE), vital sign assessments, 12- lead ECG, clinical laboratory assessments, and by general observations
11. Women of child bearing potential, must be using highly effective methods of birth control (failure rate <1% per year when used consistently and correctly) at least 4 weeks prior to Screening until Day 85. Women should be informed of the potential risks associated with becoming pregnant while enrolled. Accepted forms of contraception are implants, injectables, combined oral contraceptives, and some intrauterine devices (IUDs). In addition, a barrier method must always be used concomitantly to the highly effective method. Double-barrier is not considered a highly effective method. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) is not an acceptable means of contraception. Female patients are considered to not be of child-bearing potential when they are post-menopausal for at least 2 years with follicle-stimulating hormone (FSH) levels >40 mIU/mL, are surgically sterilized, or have undergone hysterectomy.
12. Male patients with female partners of childbearing potential must agree to use a condom without spermicide during sexual activity with female partners of childbearing potential. Female sexual partners of male patients must be willing to avoid pregnancy according to the above described methods.

Exclusion Criteria:

1. Known hypersensitivity to any constituent of the study drug
2. Presence of an associated hematologic non-mast-cell lineage disorder or MC leukemia
3. Any disease or condition (medical or surgical) which, in the opinion of the Investigator, might compromise the hematologic, cardiovascular, pulmonary, renal, gastrointestinal, hepatic, skeletal, or central nervous system; or other conditions that may interfere with the absorption, distribution, metabolism or excretion of AK002, or would place the patient at increased risk
4. The presence of abnormal laboratory values considered to be clinically significant by the Investigator
5. Participation in a concurrent interventional study with the last intervention occurring within 30 days prior to administration of study drug (90 days or 5 half-lives, whichever is longer, for biologic products)
6. Treatment with chemotherapy or radiotherapy in the preceding 6 months
7. Treatment for a clinically significant helminthic parasitic infection within 6 months of screening
8. Use during the 7 days before Screening (or 5 half-lives, whichever is longer) or expected to require the use of angiotensin converting enzyme (ACE) inhibitors or beta blockers
9. Use during the 30 days before Screening (or 5 half lives, whichever is longer) or expected to require the use of omalizumab, immunosuppressive drugs, or systemic corticosteroids with a daily dose >10 mg prednisone or equivalent
10. Vaccination with live attenuated vaccines within 30 days prior to initiation of treatment in the study, during the treatment period, or vaccination expected within 5 half-lives (4 months) of the study drug administration
11. Donation or loss of >500 mL of blood within 56 days prior to administration of study drug or donation of plasma within 7 days prior to administration of study drug
12. Has not refrained from excessive caffeine consumption (>3 cups of coffee per day or equivalent) for 48 hours prior to study drug administration and agreed to this do so throughout the inpatient period
13. Positive hepatitis serology results, except for vaccinated patients or patients with past but resolved hepatitis, at Screening
14. Positive HIV serology results at Screening
15. Any other reason that in the opinion of the Investigator or the Medical Monitor makes the patient unsuitable for enrollment
16. Patient is vulnerable (e.g., patient kept in detention)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability by evaluating Clinical laboratory parameters and adverse events assessed using the CTCAE version 4 | From study start to Day 85 or early term visit

SECONDARY OUTCOMES:
Evaluate PK of AK002 in patients with ISM | Through out the study from baseline to Day 85 or early term visit
Evaluate the change from baseline in absolute peripheral counts of eosinophils and basophils. | Through out the study from screening to Day 85 or early term visit
Evaluate the change from baseline in serum tryptase and eosinophil grande protein levels. | Through out the study from screening to Day 29 or early term visit
Measure changes form baseline in the 24-hour urine histamine metabolites. | Starting pre dose on day -1 to days 1, 3 and 4
Mastocytosis Quality of Life Questionnaire | Through out the study from screening to Day 85 or early term visit

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Maurer, MD, Principal Investigator — Department of Dermatology and Allergy, Charité - Universitätsmedizin Berlin
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided